CLINICAL TRIAL: NCT06072144
Title: Investigating the Reliability and Validity of the Smart Speed Device
Brief Title: Validity and Reliability of the Smart Speed Device
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, Associate Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2023/9
Record Dates: First submitted 2023-09-22; First posted 2023-10-10 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validity and reliability study — Test-retest method will be used to assess reliability. For this purpose, participants will be re-evaluated one week later with the Smart Speed device. For validity assessment, concurrent validity and agreement between measurements will be evaluated. Concurrent validity will be assessed by correlation analysis and agreement between measurements will be assessed by Bland Altman.

SUMMARY:
The Smart Speed device developed at Zafer Teknopark in Turkey was developed to objectively assess reaction time. The aim of this study was to evaluate the validity and reliability of the Smart Speed device in comparison with BlazePod and Nelson Reaction Test.

DETAILED DESCRIPTION:
The capacity to perceive, analyze, and react to a signal is referred to as reaction time. Reaction time is influenced by many factors such as visual and auditory factors. It is also influenced by individual factors such as age, gender, body mass index, attention and fatigue. Having reaction time within normal limits is very important for maintaining activities of daily living. BlazePod is a valid and reliable device for the assessment of reaction time. The Nelson Reaction test is also a valid and reliable test frequently used in the clinic for the assessment of reaction time due to its simple and rapid application. The Smart Speed device developed at Zafer Teknopark in Turkey was developed to objectively assess reaction time. The aim of this study was to evaluate the validity and reliability of the Smart Speed device in comparison with BlazePod and Nelson Reaction Test.

ELIGIBILITY:
Inclusion Criteria:

* Without having systemic disease
* To be able to speak Turkish language

Exclusion Criteria:

* Having a problem that affects physical performance

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be healthy young people between the ages of 18-24. All participants will be recruited from Afyonkarahisar Health Sciences University Physiotherapy and Rehabilitation Department.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Assessment of reaction time | 15 minutes
  To determine the validity and reliability of the Smart Speed device in assessing reaction time

CONTACTS AND LOCATIONS:
Overall Officials: Emel TAŞVURAN HORATA, PhD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Fatma EKEN, Afyonkarahisar, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided